CLINICAL TRIAL: NCT00070122
Title: A Phase III Trial of Modified FOLFOX6 Versus CAPOX, With Bevacizumab (NSC-704865) or Placebo, as First-Line Therapy in Patients With Previously Untreated Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy and Bevacizumab in Treating Patients With Locally Advanced, Metastatic, or Recurrent Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02556; S0303; U10CA032102 (NIH); CDR0000330000 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Capecitabine; Bevacizumab; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (oxaliplatin, leucovorin calcium, fluorouracil) (Experimental): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46-48 hours beginning on day 1. Patients are further randomized to receive bevacizumab or placebo* IV over 30-90 minutes on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. NOTE: *As of 11/15/04, placebo is no longer part of treatment plan; all patients receive bevacizumab.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Biological: bevacizumab; Drug: fluorouracil; Other: laboratory biomarker analysis
- Arm II (oxaliplatin, capecitabine) (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1and oral capecitabine on days 1-15. Patients are further randomized to receive bevacizumab or placebo* as in arm I. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity NOTE: *As of 11/15/04, placebo is no longer part of treatment plan; all patients receive bevacizumab.
  Interventions: Drug: oxaliplatin; Drug: capecitabine; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
  Arms: Arm I (oxaliplatin, leucovorin calcium, fluorouracil)
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
  Arms: Arm II (oxaliplatin, capecitabine)
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm I (oxaliplatin, leucovorin calcium, fluorouracil)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as oxaliplatin, leucovorin, fluorouracil, and capecitabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells. It is not yet known which combination chemotherapy regimen with bevacizumab works better in treating colorectal cancer. This randomized phase III trial is studying giving two different combination chemotherapy regimens together with bevacizumab and comparing how well they work in treating patients with locally advanced, metastatic, or recurrent colorectal cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare overall survival in patients with locally advanced, metastatic, or recurrent colorectal cancer treated with fluorouracil, leucovorin calcium, oxaliplatin, and bevacizumab vs capecitabine, oxaliplatin, and bevacizumab.

II. Compare progression-free survival and time to treatment failure in patients treated with these regimens.

III. Compare the response of patients with measurable disease treated with these regimens.

IV.Compare toxicity rates of these regimens in these patients. V. Compare patient-reported functional status and convenience of therapy in patients treated with these regimens.

VI. Correlate germline polymorphisms of DNA repair (e.g., ERCC-1, XRCC1, GST-P1, XPD, and ribonucleotide reductase), target enzymes (e.g., thymidylate synthase, dihydropyrimidine dehydrogenase, and thymidine phosphorylase), angiogenesis (e.g., vascular endothelial growth factor), and growth factors (e.g., epithelial growth factor receptor) with survival, progression-free survival, and toxicity from chemotherapy in patients treated with these regimens.

VII. Correlate tumor mRNA expression levels of similar DNA repair enzymes as well as enzymes involved in angiogenesis with survival and progression-free survival in patients treated with these regimens.Correlate tumor mRNA expression levels of similar target enzymes before treatment with survival, progression-free survival, and toxicity in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to Zubrod performance status (0 or 1 vs 2) and prior adjuvant therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46-48 hours beginning on day 1. Patients are further randomized to receive bevacizumab or placebo* IV over 30-90 minutes on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. NOTE: *As of 11/15/04, placebo is no longer part of treatment plan; all patients receive bevacizumab.

ARM II: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine on days 1-15. Patients are further randomized to receive bevacizumab or placebo* as in arm I. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. NOTE: *As of 11/15/04, placebo is no longer part of treatment plan; all patients receive bevacizumab.

Patients are followed every 3 months until disease progression. After disease progression, patients are followed every 6 months for 2 years and then annually for up to 4 years after study entry.

PROJECTED ACCRUAL: A total of 2,200 patients (1,100 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced, recurrent, or metastatic colorectal adenocarcinoma

  * Not curable by surgery or amenable to radiotherapy with curative intent
  * Previously resected colorectal cancer with new evidence of metastasis does not require separate histologic or cytologic confirmation unless one of the following is true:

    * More than 5 years has elapsed between primary surgery and development of metastatic disease
    * Primary tumor was T1-T2, N0, M0
* Site of primary lesion must be or have been in the large bowel as determined by endoscopy, radiology, or surgery
* Measurable or evaluable disease
* No known brain or leptomeningeal disease
* Performance status - Zubrod 0-2
* No history of hemorrhagic or thrombotic disorders
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Bilirubin no greater than 2.0 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN (5 times ULN for patients with liver involvement)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN for patients with liver involvement or 10 times ULN for patients with bone involvement)
* INR no greater than 1.5
* PTT no greater than ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 50 mL/min
* Proteinuria less than 1+*
* Protein less than 500mg/24 hours*
* No uncontrolled hypertension

  * Hypertension must be well-controlled (i.e., less than 160/90) and on a stable regimen of antihypertensive therapy
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled cardiac arrhythmia
* No New York Heart Association class III or IV heart disease
* No symptomatic pulmonary fibrosis
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* No active or uncontrolled severe infection
* No contraindication to oral medications (e.g., severe dysphagia)

  * G-tubes or J-tubes allowed
* No peripheral neuropathy greater than grade 1
* No serious non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No other severe acute or chronic medical condition or laboratory abnormality that would preclude study participation
* No psychiatric condition that would preclude study participation
* No prior bevacizumab
* No prior oxaliplatin
* No prior chemotherapy for advanced colorectal cancer

  * Prior adjuvant therapy for resected stage II-III disease allowed provided at least 12 months have elapsed between completion of therapy and diagnosis of recurrent disease
* At least 28 days since prior radiotherapy and recovered
* See Disease Characteristics
* More than 28 days since prior major surgical procedure or open biopsy
* More than 7 days since prior fine needle aspiration or core biopsy
* No concurrent major surgery
* More than 10 days since prior full-dose aspirin (325 mg)
* No concurrent antiplatelet agents (e.g., dipyridamole, ticlopidine, clopidogrel, or cilostazol)
* No other concurrent investigational agents
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation of central venous lines allowed
  * Low-dose prophylactic enoxaparin or heparin allowed
* No concurrent cimetidine
* No concurrent sorivudine or its related analogs (e.g., brivudine)
* No concurrent use of a cold cap or iced mouth rinses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2004-04; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall survival in patients with colorectal cancer treated with fluorouracil/leucovorin calcium and oxaliplatin with and without becavizumab versus those treated with capecitabine and oxaliplatin with our without bevacizumab | Up to 6 years
  Will be analyzed primarily by the stratified Cox model.

SECONDARY OUTCOMES:
Time to treatment failure | Up to 6 years
  Will be analyzed primarily by the Cox stratified model.
Progression-free survival | Up to 6 years
  Will be analyzed primarily by the Cox stratified model.
Response (among patients with measurable disease) | Up to 6 years
  Will be analyzed primarily by the Cox stratified model.
Treatment toxicities graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 3.0) | Up to the time of progression
Change in FACT-C TOI | Baseline to 25 weeks
  The analysis for evaluating this change will be a comparison of the change score between the first and last assessment. If cohort patterns for mean scores do not show signs of informative missing data, a mixed effects linear model approach will be used to measure change in FACT-C TOI scores.
Change in Chemotherapy Convenience and Satisfaction Questionnaire scores | Baseline to 25 weeks
  Effect size will be used to compare the size of the difference in each arm.
Whether gene expression variables are predictive of survival and progression-free survival | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Blanke, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States